CLINICAL TRIAL: NCT00775762
Title: Anti-Inflammatory and Anti-Platelet Effect of Clopidogrel and Aspirin vs Aspirin Alone in Symptomatic Polyvascular Disease and in Patients With Multiple Recurrent Cardiovascular Events
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Luigi Marzio Biasucci, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2008-004626-17
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Polyvascular Disease; Cardiovascular Disease
Keywords: Symptomatic Polyvascular disease; Multiple recurrent cardiovascular events
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- aspirin (Active Comparator)
  Interventions: Drug: aspirin
- clopidogrel (Active Comparator)
  Interventions: Drug: clopidogrel
- clopidogrel plus aspirin (Active Comparator)
  Interventions: Drug: clopidogrel plus aspirin

INTERVENTIONS:
Drug: aspirin — Aspirin (75-100 mg)die for three months
  Arms: aspirin
Drug: clopidogrel — Clopidogrel (75mg) die for three months
  Arms: clopidogrel
Drug: clopidogrel plus aspirin — clopidogrel 75 mg die plus aspirin 75-100 mg for three months
  Arms: clopidogrel plus aspirin

SUMMARY:
This is a monocentric, randomized, opened study to assess the anti-inflammatory and anti-platelet effect of Clopidogrel and aspirin versus aspirin or clopidogrel alone in patients with symptomatic polyvascular disease and with multiple recurrent cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic polyvascular disease or recurrent cardiovascular events. In particular patients with established stable coronary artery disease associated with peripheral disease or cerebrovascular disease and patients with more than two acute cardiovascular events.

Exclusion Criteria:

* chronic treatment with anticoagulant drugs and the use of other antiplatelet therapy;
* intolerance/allergy to Aspirin or to Clopidogrel
* platelet counts outside the range of 125-450 10^9/l
* inflammatory or infectious disease
* malignancies or immunologic or hematological disorders.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-01 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The aim of the present study is to demonstrate the superior antinflammatory effect of Clopidogrel and Aspirin vs Aspirin or Clopidogrel alone in term of levels of selected circulating inflammatory markers | three months

SECONDARY OUTCOMES:
The aim of the present study is to demonstrate the superior antiplatelet effect of Clopidogrel and Aspirin vs Aspirin or Clopidogrel alone in term of TXA2 serum levels | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Department of Cardiovascular Medicine, Rome, Italy